CLINICAL TRIAL: NCT05512520
Title: Systemic Therapy Combined With Thoracic Concurrent Chemoradiotherapy Versus Systemic Therapy Alone in Stage IVB Esophageal Squamous Cell Carcinoma: A Prospective Randomized Phase II Study
Brief Title: Concurrent Chemoradiotherapy for Stage IVB Esophageal Squamous Cell Carcinoma（EC-CRT-003）
Acronym: EC-CRT-003
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Mian XI, principal investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-FXY-040
Record Dates: First submitted 2022-08-21; First posted 2022-08-23 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Esophageal Squamous Cell Carcinoma
Keywords: metastatic esophageal squamous cell carcinoma; anti-PD-1; Capecitabine; chemoradiotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Concurrent Chemoradiotherapy group (Experimental): After completion of 4 to 6 cycles of standard chemotherapy and anti-PD1, all patients will receive thoracic radiation therapy (RT) in the following scheme: 45 to 50.4Gy in 25 to 28 fractions, concurrently with 2 cycles of capecitabine tablets (825mg/m2) for two weeks, and then followed by a maintenance treatment phase of anti-PD1 every 3 weeks.
  Interventions: Combination Product: Intensity-modulated radiotherapy concurrent with capecitabine
- Control group (No Intervention): After completion of 4 to 6 cycles of standard chemotherapy and anti-PD1, patients will receive the maintenance treatment with anti-PD1 every 3 weeks.

INTERVENTIONS:
Combination Product: Intensity-modulated radiotherapy concurrent with capecitabine — All patients received external-beam radiation using intensity-modulated radiotherapy. The prescribed dose is 45 to 50.4Gy in 25 to 28 fractions, concurrently with 2 cycles of capecitabine tablets (825mg/m2) for two weeks.
  Arms: Concurrent Chemoradiotherapy group

SUMMARY:
Retrospective studies suggested that the addition of thoracic concurrent chemoradiotherapy to systemic chemotherapy improved the survival and quality of life (QOL) of patients with metastatic esophageal squamous cell carcinoma (ESCC). However, no prospective study had been conducted to confirm these findings. Recently, immunotherapy targeting the PD-1/PD-L1 checkpoints combined with chemotherapy had been proved to significantly prolong the survival of those patients compared with chemotherapy alone. Moreover, anti-PD-1 combined with radiotherapy exerts a synergistic anti-tumor effect, which may further improve the combination efficacy. This randomized, phase II study aimed to evaluate the efficacy and safety of the chemotherapy and anti-PD-1 combined with concurrent chemoradiotherapy to primary tumor versus systemic therapy alone in stage IVB ESCC. Of note, non-regional lymph node metastasis only was the stratification factor in the random assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group performance status ≤ 2
2. Histologically confirmed squamous cell carcinoma of the esophagus;
3. Diagnosed with stage IVB disease (according to UICC TNM version 8);
4. Received 4 to 6 cycles of standard chemotherapy (fluoropyrimidine or taxane-based platinum doublet chemotherapy) and anti-PD1 treatment, and no progression disease was confirmed;
5. Estimated life expectancy >4 months;
6. The function of important organs meet the following requirements: a. white blood cell count (WBC) ≥ 4.0×109/L, absolute neutrophil count (ANC) ≥ 1.5×109/L; b. platelets ≥ 100×109/L; c. hemoglobin ≥ 9g/dL; d. serum albumin ≥ 2.8g/dL; e. total bilirubin ≤ 1.5×ULN, ALT, AST and/or AKP ≤ 2.5×ULN; f. serum creatinine ≤ 1.5×ULN or creatinine clearance rate >60 mL/min;
7. Ability to understand the study and sign informed consent.

Exclusion Criteria:

1. Progression was confirmed after completion of 4 to 6 cycles of standard chemotherapy and anti-PD1 treatment;
2. Patients with intracranial metastasis disease at diagnosis;
3. History of thoracic irradiation;
4. Known or suspected allergy or hypersensitivity to monoclonal antibodies and the chemotherapeutic drugs: Capecitabine, paclitaxel, or platinum;
5. Patients who have a preexisting esophagomediastinal fistula and/or esophagotracheal fistula;
6. A history of malignancies other than esophageal cancer before enrollment, excluding non-melanoma skin cancer, in situ cervical cancer, or cured early prostate cancer
7. Patients who cannot tolerate chemoradiotherapy due to severe cardiac, lung, liver, or kidney dysfunction, or hematopoietic disease or cachexia.
8. Inability to provide informed consent due to psychological, familial, social, and other factors;
9. Female patients who are pregnant or during lactation;
10. Active autoimmune diseases, a history of autoimmune diseases (including but not limited to these diseases or syndromes, such as colitis, hepatitis, hyperthyroidism), a history of immunodeficiency (including a positive HIV test result), or other acquired or congenital immunodeficiency diseases, a history of organ transplantation or allogeneic bone marrow transplantation;
11. A history of interstitial lung disease or non-infectious pneumonia;
12. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (positive for hepatitis C antibody, and HCV-RNA levels higher than the lower limit of the assay).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
1-year progression-free survival | From date of randomization until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 12 months
  The 1-year progression-free survival of each group

SECONDARY OUTCOMES:
1-year overall survival | From date of randomization until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 12 months
  The 1-year overall survival of the each group
ORR | 3 months after chemoradiotherapy (plus or minus 14 days)
  Overall response rate
Treatment-related adverse events | From the start of treatment to 2 year after the completion of treatment
  Toxicity of treatment was evaluated according to CTCAE 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen University Cancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guttmann DM, Mitra N, Bekelman J, Metz JM, Plastaras J, Feng W, Swisher-McClure S. Improved Overall Survival with Aggressive Primary Tumor Radiotherapy for Patients with Metastatic Esophageal Cancer. J Thorac Oncol. 2017 Jul;12(7):1131-1142. doi: 10.1016/j.jtho.2017.03.026. Epub 2017 Apr 28. PMID 28461255
- [Background] Liu S, Luo L, Zhao L, Zhu Y, Liu H, Li Q, Cai L, Hu Y, Qiu B, Zhang L, Shen J, Yang Y, Liu M, Xi M. Induction chemotherapy followed by definitive chemoradiotherapy versus chemoradiotherapy alone in esophageal squamous cell carcinoma: a randomized phase II trial. Nat Commun. 2021 Jun 29;12(1):4014. doi: 10.1038/s41467-021-24288-1. PMID 34188053